CLINICAL TRIAL: NCT01860898
Title: A Phase I Study of iPS Cell Generation From Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dennis Wigle, M.D., P.h.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09-005334
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Thoracic Diseases; Respiratory Tract Diseases; Cancer of Lung; Cancer of the Lung; Lung Cancer; Lung Diseases, Obstructive; COPD; Pulmonary Emphysema; Neoplasms, Lung; Neoplasms, Pulmonary; Pulmonary Cancer; Pulmonary Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell
Keywords: lung; cancer; thoracic; chest; pulmonary
MeSH Terms: conditions — Thoracic Diseases; Respiratory Tract Diseases; Lung Neoplasms; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive; Pulmonary Emphysema; Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin Biopsy (Other)
  Interventions: Other: Skin Biopsy

INTERVENTIONS:
Other: Skin Biopsy — Biopsy samples will be taken as a 2mm x 2cm excision of a wedge of skin at the edge of the incision during your surgery at the Mayo Clinic Rochester. Such excisions are frequently done as part of routine skin closure for optimal skin cosmesis following the surgical procedure.

SUMMARY:
As part of the long-term goal of successfully implementing tissue regeneration strategies in an individualized manner for patients with thoracic diseases including, but not limited to: cystic fibrosis, pulmonary fibrosis and pulmonary hypertension, the investigators will assess the feasibility of collecting skin biopsies from patients undergoing surgery for thoracic disease, culturing skin fibroblasts from the biopsy, and reprogramming these skin fibroblasts into induced pluripotent cells.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Thoracic Surgery at the Mayo Clinic Rochester
* Presence of a Thoracic Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-09; Primary Completion 2014-10-28 (Actual); Study Completion 2014-10-28 (Actual)

PRIMARY OUTCOMES:
Feasibility | 1 year
  As part of the long-term goal of successfully implementing tissue regeneration strategies in an individualized manner for patients with thoracic diseases including, but not limited to: cystic fibrosis, pulmonary fibrosis and pulmonary hypertension, we will assess the feasibility of collecting skin biopsies from patients undergoing surgery for thoracic disease, culturing skin fibroblasts from the biopsy, and reprogramming these skin fibroblasts into induced pluripotent cells. Markers of induced pluripotent phenotype will be utilized to assess successful reprogramming.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis A Wigle, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials